CLINICAL TRIAL: NCT02104193
Title: The Effect of Simvastatin on the Clinical Outcome of Patients With Brain Metastases Treated With Radiation Therapy: a Pilot Study
Brief Title: Simvastatin Effect on Radiation Therapy of Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, MAy Ahmed Shawki, teaching assisstant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH CL 25
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Brain Metastases
Keywords: brain metastases; simvastatin; radiation therapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Simvastatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- simvastatin (Experimental): they will receive simvastatin in addition to radiation therapy
  Interventions: Drug: simvastatin in addition to radiation therapy
- control (Active Comparator): they will receive radiation therapy only
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Drug: simvastatin in addition to radiation therapy — simvastatin 80 mg tablet once daily during the radiation therapy period in addition to radiation therapy 30 Gy delivered in 10 fractions over 2 weeks
  Arms: simvastatin
Radiation: radiation therapy — radiation therapy 30 Gy delivered in 10 fractions over 2 weeks
  Arms: control

SUMMARY:
The purpose of the study is to evaluate the effect of simvastatin in combination with radiotherapy on the clinical outcomes of patients with brain metastases.

DETAILED DESCRIPTION:
Despite current advances in therapies, the outcome for patients with brain metastases is fatal. New therapeutic approaches, such as radiosensitizing agents, are needed to provide a significant survival advantage for those patients. Statins have been reported to enhance the efficacy of radiotherapy in addition to a neuroprotective effect. The aim of the study is to evaluate the effect of simvastatin on the efficacy and safety of radiation therapy in patients with brain metastases and on improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable brain metastases
* Age more than 18 years old
* Patients should be planned for radiation therapy

Exclusion Criteria:

* Renal dysfunction (more than 1 upper normal level)
* Hepatic dysfunction (alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3 times the upper normal level )
* Pregnancy or lactation.
* Known hypersensitivity to simvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
a- Response rate | 4 weeks after radiation therapy
  brain CT/MRI will be done at baseline and 4 weeks after radiotherapy to evaluate the reduction in tumor size

SECONDARY OUTCOMES:
progression free and overall survival | up to 6 months
  it measures time from treatment initiation to either progression or death from any cause
adverse effects | during the treatment period
  any adverse/side effect will be evaluated

OTHER OUTCOMES:
quality of life | baseline, after radiation therapy, 6 weeks, 18 weeks, 30 weeks
  measures the patient quality of life
cognitive function assessment using Montreal cognitive assessment test | baseline, after radiation therapy, 6 weeks, 18 weeks, 30 weeks
  assess the patient cognitive function by the evaluation of Montreal cognitive assessment test score
serum s100 B protein | baseline, after radiation therapy
  evaluate serum s100 B protein at baseline and after 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: May A Shawki, master, Principal Investigator — Faculty of Pharmacy- Ain Shams university
Locations (1):
- Ain Shams university Hospitals, Cairo, Egypt